CLINICAL TRIAL: NCT06231082
Title: Bloody or Well Done. How Would You Like Your Liver Biopsy, Sir? Post Liver bIopsy abdoMinal PaIn as Predictive Factor for Liver bleeDing (LIMPID)
Brief Title: Bloody or Well Done. How Would You Like Your Liver Biopsy, Sir?
Acronym: LIMPID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, Associate Professor of Gastroenterology, Carol Davila University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LIMPID
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Liver Disease Parenchymal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group one - percutaneous (P) (Active Comparator): Percutaneous procedure will be performed under standard conditions, under transabdominal ultrasound guidance. After choosing the optimum needle trajectory, the skin site will be marked, standard skin sterilization with iodine and surgical draping of the site will be performed. Local anesthesia of the site with gradual lidocaine solution infiltration of the skin and underlying planes will be performed. Under ultrasound guidance, with collaboration of the patient for the respiratory movements, one or two passages with a 16G needle will be performed (BARD Max Core 16G, Becton Dickinson, USA). Specimens will be collected in formalin and send to pathology for processing.
  Interventions: Procedure: Group one - percutaneous (P)
- Group two - EUS FNB (E) (Active Comparator): EUS guided liver FNB will be performed under deep sedation with propofol under anesthesiology monitoring. A 19G gauge Franseen needle (Acquire 19G, Boston Scientific, USA) will be used with the "wet suction" technique. Before inserting into the operating channel, the stylet will be removed, and the needle will be primed with heparin (500UI/5ml). After liver puncture, the 20ml aspiration syringe will be attached. Three needle actuations will be performed, one or two passes in the left liver lobe. At the end of the 3rd actuation, the syringe aspiration will be stopped, the needle will be left in place in the liver parenchyma for 2 to 3 minutes. The liver needle path will be examined with Doppler ultrasound to look for possible bleeding. If present, about 25% of the needle content will be pushed in the liver path, as previously described - the "blood patch" technique
  Interventions: Procedure: Group two - EUS FNB (E)

INTERVENTIONS:
Procedure: Group one - percutaneous (P) — Percutaneous procedure will be performed under standard conditions, under transabdominal ultrasound guidance. After choosing the optimum needle trajectory, the skin site will be marked, standard skin sterilization with iodine and surgical draping of the site will be performed. Local anesthesia of the site with gradual lidocaine solution infiltration of the skin and underlying planes will be performed. Under ultrasound guidance, with collaboration of the patient for the respiratory movements, one or two passages with a 16G needle will be performed (BARD Max Core 16G, Becton Dickinson, USA). Specimens will be collected in formalin and send to pathology for processing.
  Arms: Group one - percutaneous (P)
Procedure: Group two - EUS FNB (E) — EUS guided liver FNB will be performed under deep sedation with propofol under anesthesiology monitoring. A 19G gauge Franseen needle (Acquire 19G, Boston Scientific, USA) will be used with the "wet suction" technique. Before inserting into the operating channel, the stylet will be removed, and the needle will be primed with heparin (500UI/5ml). After liver puncture, the 20ml aspiration syringe will be attached. Three needle actuations will be performed, one or two passes in the left liver lobe. At the end of the 3rd actuation, the syringe aspiration will be stopped, the needle will be left in place in the liver parenchyma for 2 to 3 minutes. The liver needle path will be examined with Doppler ultrasound to look for possible bleeding. If present, about 25% of the needle content will be pushed in the liver path, as previously described - the "blood patch" technique.
  Arms: Group two - EUS FNB (E)

SUMMARY:
This is a randomized comparative trial between percutaneous liver biopsy and EUS FNB guided liver biopsy in patients with parenchymal liver disease.

Studies so far have been shown that EUS FNB guided liver biopsy is non inferior to percutaneous liver biopsy in terms of efficacy, provided several conditions are met (type of needle, wet suction, actuations).

În terms of safety, it may be that EUS FNB have an advantage, as needle diameter is slightly smaller, needle is inserted under better visualisation especially in patients with large subcutaneous fat tissue and the possibility of examining the needle tract and plugging it with needle content if needed ("the blood patch technique").

However, although severe, the incidence of liver bleeding is low, so a comparative trial with the hypothesis that EUS FNB has fewer liver bleedings than percutaneous techniques would have a very large sample size.

A recent study found out that abdominal pain at 2 hours after procedure is predictive for liver bleeding.

So we have design a randomized prospective trial assuming that EUS FNB guided liver biopsy has significantly less abdominal pain at 2 hours after procedure when compared to percutaneous route, using abdominal pain at 2 hours as a surrogate marker for risk of liver bleeding.

DETAILED DESCRIPTION:
Why liver biopsy? Parenchymal liver diseases need sometimes diagnostic or staging assessment liver biopsy (eg. autoimmune hepatitis, primary biliary cholangitis, metabolic dysfunction associated fatty liver disease - MAFLD). Also, some focal liver lesions may need a diagnostic liver biopsy (eg. primitive liver tumors, liver metastases).

This can be performed percutaneously, trans-jugular and more recently trans-gastric or trans-duodenal under endoscopic ultrasound (EUS) guidance. The trans-jugular route was proposed for patients with coagulation disorders, as there is virtually no risk of bleeding, as the procedure is done within the supra-hepatic veins.

Currently, evidence exist that optimal results for EUS guided fine needle biopsy (FNB) are obtained by using a 19 Gauge Franseen FNB needle, by the heparin primed "wet suction" technique, with one or two passes (in both liver lobes), with at least 3 needle actuations [1,2,3,4]. Ensuring these conditions, the outcomes are non-inferior to percutaneous liver biopsy (length of the specimen, number of portal tracts, diagnostic accuracy).

So why choose EUS guided liver FNB? Two percutaneous liver biopsy adverse reactions are probably responsible for one's apprehension towards it - post procedure abdominal pain and the risk of liver bleeding. A recent meta-analysis [5] has found an incidence of mild abdominal pain at 12.9% and moderate-severe abdominal pain at 0.34%. The percentages for liver bleeding were 0.48% for major bleeding, 0.11% for major hematoma, 0.06% for hemoperitoneum and 0.01% for haemobilia (0.66% in total).

Bisonnette et al [6] have tried to find predictive factors for liver bleeding after percutaneous or trans-jugular liver biopsy. The only predictive factor was pain at 2h liver biopsy. This was more frequent following percutaneous than trans-jugular liver biopsy (33% vs. 15%; p < .001). Out of all patients with pain 2 h after liver biopsy, 15% had a liver biopsy-related bleeding, while out of those without pain 2 h after liver biopsy, 4% had a liver biopsy-related bleeding (p = .002). Pain 2 h after liver biopsy had a 55% (95% CI 0.35-0.73) sensitivity, 75% (95% CI 0.70-0.80) specificity, and 96% (95% CI 0.93-0.97) negative predictive value for liver biopsy -related bleeding.

EUS guided liver FNB seems to be safer than percutaneous liver biopsy. Eleven studies so far on 632 patients who had EUS FNB with 19G Franseen needle report on post procedure liver bleeding and abdominal pain [7-17]. Abdominal pain was present in 7.7%. of cases (28 of 362 reported patients), while liver bleeding was present in 0.16% (1 of 593, as "bile leak").

If we we're to design a study to prove that EUS guided liver FNB decreases bleeding rate from 0.66% for percutaneous route to 0.16%, with a type I error probability of 5% and a power of 80%, we would need to include 5126 patients, that is 2563 for each arm in a 1:1 allocation [7]. This is a near impossible study.

However, as Bisonnette et al [6] have proven, pain at 2h after liver biopsy is predictive for liver bleeding. So, we only need to prove that EUS guided liver FNB significantly decreases abdominal pain at 2h after procedure as compared to percutaneous route.

So, to prove that EUS guided liver FNB decreases abdominal pain rate at 2h after biopsy from 33% for percutaneous method to 7.7%, with a type I error probability of 5% and a power of 80%, we would need to include 78 patients, that is 39 for each arm in a 1:1 allocation [7].

Question of the research project We aim to answer the question whether EUS guided liver FNB has a significantly lower rate of abdominal pain at 2h after procedure than percutaneous liver biopsy.

Hypothesis The EUS guided liver FNB has a significantly lower rate of abdominal pain at 2h after procedure than percutaneous liver biopsy, which probably translates in a significantly lower liver bleeding rate.

Patients will be randomly allocated in one of the 2 study groups, following a randomization list (www.random.org), as it follows:

* Group one - percutaneous (P)
* Group two - EUS FNB (E)

Group one (P) - Percutaneous procedure will be performed under standard conditions, under transabdominal ultrasound guidance. After choosing the optimum needle trajectory, the skin site will be marked, standard skin sterilization with iodine and surgical draping of the site will be performed. Local anesthesia of the site with gradual lidocaine solution infiltration of the skin and underlying planes will be performed. Under ultrasound guidance, with collaboration of the patient for the respiratory movements, one or two passages with a 16G needle will be performed (BARD Max Core 16G, Becton Dickinson, USA). Specimens will be collected in formalin and send to pathology for processing.

Group two (E) - EUS guided liver FNB will be performed under deep sedation with propofol under anesthesiology monitoring. A 19G gauge Franseen needle (Acquire 19G, Boston Scientific, USA) will be used with the "wet suction" technique. Before inserting into the operating channel, the stylet will be removed, and the needle will be primed with heparin (500UI/5ml). After liver puncture, the 20ml aspiration syringe will be attached. Three needle actuations will be performed, one or two passes in the left liver lobe. At the end of the 3rd actuation, the syringe aspiration will be stopped, the needle will be left in place in the liver parenchyma for 2 to 3 minutes. The liver needle path will be examined with Doppler ultrasound to look for possible bleeding. If present, about 25% of the needle content will be pushed in the liver path, as previously described - the "blood patch" technique [19].

ELIGIBILITY:
Inclusion Criteria:

* Diffuse parenchymal liver disease with indication for liver biopsy for diagnostic and/or staging purposes,
* Eligibility for deep sedation with propofol
* Age above 18 years old
* Informed consent

Exclusion Criteria:

* Coagulation disorders which cannot be corrected
* Anticoagulant and/or antiagregant medication which cannot be stopped temporarily.
* Contraindications for liver biopsy, to local lidocaine anesthesia and to deep propofol sedation
* Absence of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Post procedure pain at 2 hours after procedure | 2 hours
  Post procedure pain at 2 hours measured by Visual Analogue Scale (0 - 10)

SECONDARY OUTCOMES:
Post procedure pain at 24 hours after procedure | 24 hours
  Post procedure pain at 24 hours measured by Visual Analogue Scale (0 - 10)
Proportion of post procedure liver bleeding | 7 days
  Proportion of post procedure liver bleeding = number of patients with (perihepatic fluid, hemoperitoneum, liver hematoma, hemorrhagic shock) divided by the total number of patients enrolled in one arm
Longest intact specimen | 2 hours
  Length (mm) of the longest intact specimen removed by biopsy for one patient
Aggregate specimen length | 2 hours
  Sum of the length of all the specimens (mm) removed by biopsy for one patient
Total number of specimens | 2 hours
  Sum of the number of specimens removed by biopsy for one patient
Proportion of specimens > 20mm in aggregate length | 2 hours
  Proportion of specimens > 20mm in aggregate length = number of patients with aggregate length of specimens (secondary outcome 5) > 20mm divided by the total number of patients enrolled in one arm
Total specimen complete portal tracts (CPT) | 28 days
  Sum of CPT for all specimens removed by biopsy for one patient
Proportion of specimens with > 11 CPT | 28 days
  Proportion of specimens with > 11 CPT = number of patients with specimens > 11 CPT divided by the total number of patients in each arm
Proportion of specimen with conclusive pathological diagnosis | 28 days
  Proportion of specimen with conclusive pathological diagnosis = number of patients with conclusive pathological diagnosis divided by the total number of patients in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- "Prof. Dr. Agrippa Ionescu" Clinical and Emerency Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Facciorusso A, Crino SF, Ramai D, Fabbri C, Mangiavillano B, Lisotti A, Muscatiello N, Cotsoglou C, Fusaroli P. Diagnostic yield of endoscopic ultrasound-guided liver biopsy in comparison to percutaneous liver biopsy: a systematic review and meta-analysis. Expert Rev Gastroenterol Hepatol. 2022 Jan;16(1):51-57. doi: 10.1080/17474124.2022.2020645. Epub 2021 Dec 29. PMID 34918578
- [Background] Zeng K, Jiang Z, Yang J, Chen K, Lu Q. Role of endoscopic ultrasound-guided liver biopsy: a meta-analysis. Scand J Gastroenterol. 2022 May;57(5):545-557. doi: 10.1080/00365521.2021.2025420. Epub 2022 Jan 20. PMID 35049405
- [Background] Chandan S, Deliwala S, Khan SR, Mohan BP, Dhindsa BS, Bapaye J, Goyal H, Kassab LL, Kamal F, Sayles HR, Kochhar GS, Adler DG. EUS-guided versus percutaneous liver biopsy: A comprehensive review and meta-analysis of outcomes. Endosc Ultrasound. 2023 Mar-Apr;12(2):171-180. doi: 10.4103/EUS-D-21-00268. PMID 36204798
- [Background] Laleman W, Vanderschueren E, Mehdi ZS, Wiest R, Cardenas A, Trebicka J. Endoscopic procedures in hepatology: Current trends and new developments. J Hepatol. 2024 Jan;80(1):124-139. doi: 10.1016/j.jhep.2023.08.032. Epub 2023 Sep 18. PMID 37730125
- [Background] Thomaides-Brears HB, Alkhouri N, Allende D, Harisinghani M, Noureddin M, Reau NS, French M, Pantoja C, Mouchti S, Cryer DRH. Incidence of Complications from Percutaneous Biopsy in Chronic Liver Disease: A Systematic Review and Meta-Analysis. Dig Dis Sci. 2022 Jul;67(7):3366-3394. doi: 10.1007/s10620-021-07089-w. Epub 2021 Jun 15. PMID 34129125
- [Background] Bissonnette J, Riescher-Tuczkiewicz A, Gigante E, Bourdin C, Boudaoud L, Soliman H, Durand F, Ronot M, Valla D, Vilgrain V, de Raucourt E, Rautou PE. Predicting bleeding after liver biopsy using comprehensive clinical and laboratory investigations: A prospective analysis of 302 procedures. J Thromb Haemost. 2022 Dec;20(12):2786-2796. doi: 10.1111/jth.15888. Epub 2022 Oct 5. PMID 36128757
- [Background] Ching-Companioni RA, Diehl DL, Johal AS, Confer BD, Khara HS. 19 G aspiration needle versus 19 G core biopsy needle for endoscopic ultrasound-guided liver biopsy: a prospective randomized trial. Endoscopy. 2019 Nov;51(11):1059-1065. doi: 10.1055/a-0956-6922. Epub 2019 Jul 23. PMID 31342474
- [Background] Nieto J, Dawod E, Deshmukh A, Penn E, Adler D, Saab S. EUS-guided fine-needle core liver biopsy with a modified one-pass, one-actuation wet suction technique comparing two types of EUS core needles. Endosc Int Open. 2020 Jul;8(7):E938-E943. doi: 10.1055/a-1165-1767. Epub 2020 Jun 16. PMID 32617398
- [Background] Aggarwal SN, Magdaleno T, Klocksieben F, MacFarlan JE, Goonewardene S, Zator Z, Shah S, Shah HN. A prospective, head-to-head comparison of 2 EUS-guided liver biopsy needles in vivo. Gastrointest Endosc. 2021 May;93(5):1133-1138. doi: 10.1016/j.gie.2020.09.050. Epub 2020 Oct 9. PMID 33045222
- [Background] Ching-Companioni RA, Johal AS, Confer BD, Forster E, Khara HS, Diehl DL. Single-pass 1-needle actuation versus single-pass 3-needle actuation technique for EUS-guided liver biopsy sampling: a randomized prospective trial (with video). Gastrointest Endosc. 2021 Sep;94(3):551-558. doi: 10.1016/j.gie.2021.03.023. Epub 2021 Mar 23. PMID 33771557
- [Background] Bang JY, Ward TJ, Guirguis S, Krall K, Contreras F, Jhala N, Navaneethan U, Hawes RH, Varadarajulu S. Radiology-guided percutaneous approach is superior to EUS for performing liver biopsies. Gut. 2021 Dec;70(12):2224-2226. doi: 10.1136/gutjnl-2021-324495. Epub 2021 Mar 25. No abstract available. PMID 33766911
- [Background] Hashimoto R, Lee DP, Samarasena JB, Chandan VS, Guo W, Lee JG, Chang KJ. Comparison of Two Specialized Histology Needles for Endoscopic Ultrasound (EUS)-Guided Liver Biopsy: A Pilot Study. Dig Dis Sci. 2021 May;66(5):1700-1706. doi: 10.1007/s10620-020-06391-3. Epub 2020 Jun 17. PMID 32556821
- [Background] Ali AH, Nallapeta NS, Yousaf MN, Petroski GF, Sharma N, Rao DS, Yin F, Davis RM, Bhat A, Swi AIA, Al-Juboori A, Ibdah JA, Hammoud GM. EUS-guided versus percutaneous liver biopsy: A prospective randomized clinical trial. Endosc Ultrasound. 2023 May-Jun;12(3):334-341. doi: 10.1097/eus.0000000000000010. Epub 2023 Jul 25. PMID 37693114
- [Background] Choi AY, Li X, Guo W, Chandan VS, Samarasena J, Lee JG, Chang KJ, Hu KQ. Performance of Endoscopic Ultrasound-Guided Versus Percutaneous Liver Biopsy in Diagnosing Stage 3-4 Fibrosis. Dig Dis Sci. 2023 Sep;68(9):3774-3780. doi: 10.1007/s10620-023-08019-8. Epub 2023 Aug 4. PMID 37540389
- [Background] Rai P, Majeed A, Kumar P, Rajput M, Goel A, Rao RN. Endoscopic ultrasound-guided liver biopsy using a single-pass, slow-pull technique with a 19-G Franseen tip fine-needle biopsy needle: A prospective study. Indian J Gastroenterol. 2023 Jun;42(3):418-424. doi: 10.1007/s12664-023-01339-7. Epub 2023 Apr 25. PMID 37097513
- [Background] Sundaram S, Shah B, Jagtap N, Angadi S, Jain AK, Afzalpurkar S, Giri S. Diagnostic efficacy of endoscopic ultrasound-guided liver biopsy for diffuse liver diseases and its predictors - a multicentric retrospective analysis. Clin Exp Hepatol. 2023 Sep;9(3):243-250. doi: 10.5114/ceh.2023.130618. Epub 2023 Aug 23. PMID 37790688
- [Background] Sowa P, Kolb J, Samarasena J, Chang KJ. EUS-guided blood patch delivery during liver biopsy: nature's gel foam. VideoGIE. 2021 Jul 22;6(11):487-488. doi: 10.1016/j.vgie.2021.06.006. eCollection 2021 Nov. PMID 34765837
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014